CLINICAL TRIAL: NCT06592690
Title: Effect of Rate-responsive Compared to VDD Pacing in Cardiac Resynchronization Therapy Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale Centrale Bolzano (Other)
Responsible Party: Principal Investigator, Luca Donazzan, Cardiologist, Ospedale Centrale Bolzano
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0100843-BZ
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Heart Failure, Wide QRS Complex
Keywords: atrial pacing; cardiac resynchronization therapy; heart failure; implantable cardioverter defibrillator; rate-adaptive pacing
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Randomized, cross-over, double-blind, multicenter study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VDD (Active Comparator): A pacing mode which allows sensing of intrinsic sinus rhythm as much as possible to avoid unnecessary atrial pacing is the preferred programming in patients with CRT without atrial pacing indication. VDD pacing mode met these criteria.
  Interventions: Other: Atrial tracking pacing mode
- DDDR (Experimental): DDDR pacing mode added atrial support to these using an accelerometer-based rate-responsive sensor which should be able to increase heart rate when needed.
  Interventions: Other: Atrial pacing support

INTERVENTIONS:
Other: Atrial pacing support — Use a pacing mode with atrial pacing including a rate-resposive sensor.
  Arms: DDDR
Other: Atrial tracking pacing mode — A pacing mode which allows sensing of intrinsic sinus rhythm as much as possible to avoid unnecessary atrial pacing is the preferred programming in patients with CRT without atrial pacing indication. VDD pacing mode met these criteria.
  Arms: VDD

SUMMARY:
This study aims to understand the best programming pacing mode for cardiac resynchronization therapy devices used to treat chronic heart failure.

DETAILED DESCRIPTION:
Cardiac resynchronization therapy (CRT) efficacy trials to date used atrial-synchronous biventricular pacing wherein there is no or minimal atrial pacing. However, bradycardia and chronotropic incompetence are common in this patient population.

Despite neutral results on hard clinical outcomes of the atrial support in CRT patients, it is not clear if a rate-responsive pacing may add incremental benefits on exercise capability.

The aim of this study is to assess the impact of RR pacing compare to VVD pacing in patients implanted with CRT devices in term of functional capacity, measured by the six-minute walking test (6MWT). This simple test has shown to be an independent predictors of mortality in this cohort of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients willing to participate in the study and signing the approved Patient Informed Consent (PIC) Form;
* Patients with approved indication for CRT by European Society of Cardiology/European Heart Rhythm Association guidelines (ESC/EHRA).
* Sinus rhythm at the time of CRT device implantation with heart rate at rest above 50 bpm.

Exclusion Criteria:

* Permanent Atrial Fibrillation;
* Inability to perform 6MWT;
* Suboptimal HF drug therapy;
* Heart rate at rest above 50 bpm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2021-09-17 (Actual); Study Completion 2021-09-17 (Actual)

PRIMARY OUTCOMES:
distance walked during the 6MWT | A consecutive 6-month treatment period with the same pacing mode.
  distance walked during the 6-minute-walking-test (6MWT)

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Centrale di Bolzano, Bolzano, Italy

IPD SHARING:
Plan to Share IPD: No
Privacy concerns.

REFERENCES:
- [Derived] Donazzan L, Bulian F, Maines M, Erckert M, Peruzza F, Rauhe WG, Giacopelli D, Manfrin M. Effect of rate-adaptive atrial support compared to VDD pacing in cardiac resynchronization therapy recipients: A randomized cross-over study. Am Heart J. 2025 Mar;281:149-156. doi: 10.1016/j.ahj.2024.12.005. Epub 2024 Dec 17. PMID 39701488